CLINICAL TRIAL: NCT04782401
Title: Comparison of the Effects of Ultrasound Guided Genicular Nerve Block Versus Physical Therapy for Knee Osteoarthritis
Brief Title: The Effects of Ultrasound Guided Genicular Nerve Block for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turkish League Against Rheumatism (Other)
Responsible Party: Principal Investigator, Dr. Elif becenen, Principal investigator, Turkish League Against Rheumatism
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRASD-TG-GB
Record Dates: First submitted 2021-02-19; First posted 2021-03-04 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genicular Nerve Block (Active Comparator)
  Interventions: Other: Ultrasound guided genicular nerve block + exercise treatment
- Physical Therapy (Active Comparator)
  Interventions: Device: Physical therapy + exercise treatment

INTERVENTIONS:
Other: Ultrasound guided genicular nerve block + exercise treatment — This method was used to inject a total of 6 mL of lidocaine plus 40 mg of triamcinolone (TA) at 3 separate target sites: the superior lateral, superior medial, and inferior medial genicular nerves plus exercise treatment
  Arms: Genicular Nerve Block
Device: Physical therapy + exercise treatment — Ten sessions of hotpack as a surface warmer, TENS as a analgezic current, ultrasound therapy as a deep warmer and exercise treatment.
  Arms: Physical Therapy

SUMMARY:
Goal: Comparison of the effects of genicular nerve block with usg and physical therapy on pain, physical function for patients with knee osteoarthritis.

Material and Methods:102 patients with osteoarthritis of the knee with Kellgren-Lawrence (K-L) class 2 or 3 were included in the study.Patients were randomized to two groups, first being injected a total of 6 mL of lidocaine plus 40 mg of triamcinolone (TA) at 3 separate target sites: the superior lateral, superior medial, and inferior medial genicular nerves with exercise treatment and second being ten sessions of hotpack as a surface warmer, TENS as a analgezic current, ultrasound therapy as a deep warmer with exercise treatment.For the first group, the ultrasound we used: 12 MHz linear transducer. (Logic E9-GE, USA).The transducer was first placed parallel to the long bone shaft and moved up or down to identify the epicondyle of the long bone. The genicular arteries were identified near the periosteal areas, which are the junctions of the epicondyle and the shafts of the femur and tibia, and confirmed by color Doppler ultrasound.Accordingly, GNB target points should be next to each genicular artery because the superior lateral, superior medial, and inferior medial genicular artery traveled along each genicular nerve. , Visual Analogue Scale for pain(VAS) was primer outcome measurement, Western Ontorio and McMaster Universities Osteoarthritis Index (WOMAC) and six minute walk tests were seconder outcome measurements of the study applied before, after (two weeks) and 12th weeks of treatment. Primer endpoint of the study is decrease at least 40% in VAS values at 2nd week, second endpoint is the improvement in the womac and 6-minute walk test observed in the 2nd week continues until the 12th week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee osteoarthritis according to the 1986 American College of Rheumatology (ACR) criteria and were in Kellgren-Lawrence (KL) Grade 2-3
* Being between the ages of 45-65

Exclusion Criteria:

* Severe knee trauma history within the six month
* Previous intraarticular hyaluronic acid or steroid injection
* Previous use of oral glucosamine
* Meniscal or connective tissue damage
* Those receiving physical therapy within the six month for knee pain
* History of inflamatuary romatologic disease
* Pregnancy and breastfeeding
* Malignancy
* Psychiatric disease
* Those with a pacemaker

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) score | Pre-intervention, Change from Baseline visual analog scale at 12th weeks
  A scale for the use of measuring pain. Minimum score of the scale is 0 and maximum is 10. Higher scores mean worse outcomes.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score | Pre-intervention, Change from baseline WOMAC score at 12th weeks
  WOMAC is a scale to assess disease-related functional status and disability. It consists of three parts with 24 simple questions in total. Five questions are related to pain (WOMAC-A), two questions to morning stiffness (WOMAC-B), and the remaining 17 questions to physical condition (WOMAC-C). Each question is scored using 4-point Likert scale (0= None, 1= Mild, 2= Moderate, 3= Severe, 4= Very severe). Higher scores indicate severe pain, increased stiffness, and functional failure. Minimum score of the scale is 0 and maximum is 100. Higher scores mean worse outcomes.
Six minute walk test | Pre-intervention, Change from baseline six minute walk test at 12th weeks
  It is an objective method to evaluate exercise tolerance. It was performed on an unobstructed bare 30 meters (m) floor where every 3 meters were marked. The patients were allowed to complete the test by reducing their walking speed or stopping and getting some rest, if needed. Maximum walking distance (meters) within six min was measured. Higher distance means better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guler T, Yurdakul FG, Onder ME, Erdogan F, Yavuz K, Becenen E, Uckun A, Bodur H. Ultrasound-guided genicular nerve block versus physical therapy for chronic knee osteoarthritis: a prospective randomised study. Rheumatol Int. 2022 Apr;42(4):591-600. doi: 10.1007/s00296-022-05101-8. Epub 2022 Feb 14. PMID 35165769